CLINICAL TRIAL: NCT02428894
Title: Characterization of the Plasma Proteome Following Left Ventricular Assist Device Implantation
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 14-1376; 14GRNT20380495 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2015-04-17; First posted 2015-04-29 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Ventricular Dysfunction, Left
MeSH Terms: conditions — Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Change in plasma proteins. [Time Frame, Days 7, 14, 30, 60, 90, and 180 post-LVAD implantation][Designated as safety issue: No]
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- LVAD recipients
  Interventions: Device: LVAD

INTERVENTIONS:
Device: LVAD
  Other Names: HeartMate II

SUMMARY:
The purpose of this study is to characterize changes in the plasma proteome over time following left ventricular assist device (LVAD) implantation.

ELIGIBILITY:
Inclusion Criteria:

* Planned HeartMate II LVAD implantation
* Planned warfarin (goal INR, 2.0-3.0) and low-dose aspirin therapy post-LVAD placement

Exclusion Criteria:

* Prior history of mechanical circulatory support;
* Body weight < 110 lbs;
* Pre-existing hemolytic, bleeding, or immunologic disorders prior to LVAD implantation;
* Severe aortic stenosis;
* Renal failure requiring dialysis;
* Hepatic dysfunction resulting in severe coagulopathies;
* Recent serious infection;
* Current need for prolonged ventilatory support;
* Prior organ transplantation;
* Blood transfusion within 14 days of the first planned study blood draw;
* Concomitant immunosuppressant or chemotherapeutic agents;
* Pregnant women;
* Decisionally challenged or prisoners;
* Unwilling to provide written informed consent

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited from the University of Colorado Hospital Advanced Heart Failure Program.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-10; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Quantitative differences in plasma protein abundance | Days 7, 14, 30, 60, 90, and 180 post-LVAD implantation

CONTACTS AND LOCATIONS:
Overall Officials: Christina Aquilante, Pharm.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States